CLINICAL TRIAL: NCT01606930
Title: A Pilot Study to Improve Patient-Doctor Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Patrick G. O'Malley, MD, MPH, Professor of Medicine, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A-14352.4
Record Dates: First submitted 2012-04-18; First posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Disease; Hypertension; Hyperlipidemia; Diabetes Mellitus; Osteoarthritis; COPD; Cardiovascular Disease
Keywords: Patient Satisfaction; Patient Doctor Communication; Shared Decision Making; Patient Activation
MeSH Terms: conditions — Chronic Disease; Hypertension; Hyperlipidemias; Diabetes Mellitus; Osteoarthritis; Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Patient Satisfaction; Patient Participation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Group (No Intervention): Group will see their physician without receiving the "activation" instrument.
- "Activated" Group (Active Comparator): Group will be given an "activation" instrument to complete before their appointment and instructed to refer to and use the instrument during their clinical encounter.
  Interventions: Behavioral: Patient Primer Tool

INTERVENTIONS:
Behavioral: Patient Primer Tool — The instrument is completed before the scheduled appointment and is designed to prompt patients to reflect on their specific goals for the medical encounter, prioritize those goals, and to "Prime" them to engage in a discussion centered on their concerns and expectations. In addition, participants will be encouraged to bring this form into their physician visit and use it to engage their clinician in a discussion about their health needs.
  Other Names: Patient Activation Tool
  Arms: "Activated" Group

SUMMARY:
The purpose of this controlled pilot study is to determine whether an intervention aimed at patients will improve partnering, shared decision-making and open communication. Results from this pilot study will inform how to best proceed with a larger multi-centered randomized controlled trial.

The specific hypothesis for this pilot study is to:

1. Test the feasibility of a simple patient-centered intervention.
2. Test the correlation between patient readiness to actively engage in conversation (assessed using a pre-visit patient survey) and actual patient behaviors in the encounter.
3. Develop a coding tool that will quantify patient activation in clinical encounters.
4. Test whether activating patients who are more involved and revealing in the patient-clinician dyad will improve patient and clinician outcomes.

DETAILED DESCRIPTION:
Chronic illness requires a greater participation by the patient in the management of their own disease process. Patients now increasingly find themselves dealing with multiple illnesses over the span of their lifetime.

Patient-provider communication is key to optimal patient outcomes. Numerous studies have shown adverse effects of poor communication on a number of outcomes, including patient and provider satisfaction as well as medical compliance and health related outcomes.

An important next step in this field is to study whether it is possible to improve chronic illness care in real world settings by improving the quality of patient-provider interaction through feasible interventions focused on efficient, motivational, and empathic communication, targeted at both patients and providers.

There is little information on the best patterns of communication in dealing with patients with multiple comorbidities. The investigators believe that an optimal healing relationship between these patients and their healthcare providers includes shared decision-making, partnering between patients and clinicians to foster health and healthy behaviors in an environment of trust, and effective open communication.

An important outcome for this pilot study is feasibility. The investigators intend to conduct a follow-up multi-centered trial; planning and budgeting for such a trial will require information gleaned from this study. What is the rate of accrual and how many patients can realistically be enrolled and followed within the current study personnel. What outcomes are sensitive to change and how much change can the investigators expect to see? Will this intervention effect change in patient behavior? This study will give us insight to allow us to build a right-sized project.

ELIGIBILITY:
Inclusion Criteria:

* Military health care beneficiaries presenting for chronic medical care with their primary care clinician
* Over the age of 18
* At least 2 and no more than 10 visits with their primary care provider in the previous year
* Receiving pharmacological treatment for hypertension
* At least 2 of the following common chronic illnesses: hyperlipidemia, chronic obstructive pulmonary disease, asthma, congestive heart failure, chronic pain, ischemic heart disease, osteoarthritis, depression, back pain, chronic headaches, or diabetes

Exclusion Criteria:

* Over the age of 80
* Incapable of completing the questionnaires, either due to cognitive impairment or lack of English-literacy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Degree of shared medical decision-making | Baseline
  Assessed from transcribed audio-tapes of the doctor-patient encounter using Roter Interaction Analysis System (RIAS).
Adherence to anti-hypertensive drug treatment at baseline | Baseline
  This outcome will be assessed using pill counts by the pharmacists.
Adherence to anti-hypertensive drug treatment at one month | One month
  This outcome will be assessed using pill counts by the pharmacists.
Adherence to anti-hypertensive drug treatment at three months | Three months
  This outcome will be assessed using pill counts by the pharmacists.

SECONDARY OUTCOMES:
Patient satisfaction | Baseline
  Post-encounter survey using the validated Rand-9 Patient Satisfaction Tool
Clinician rating of patient as "difficult" | Baseline
  Clinician Rating of the Encounter Using the Difficult Doctor-Patient Relationship Questionaire (DDPRQ).
Patient Trust in their physician at baseline | Baseline
  Validated Trust in Physician (11-item) Instrument
Patient Trust in their physician at one month | one month
  Validated Trust in Physician (11-item) Instrument
Patient Trust in their physician at three months | Three months
  Validated Trust in Physician (11-item) Instrument
Systolic and Diastolic Blood Pressure at baseline | Baseline
  Each blood pressure data point was the average of 3 measurements measured 5 minutes apart while seated.
Systolic and Diastolic Blood Pressure at one month | One month
  Each blood pressure data point was the average of 3 measurements measured 5 minutes apart while seated.
Systolic and Diastolic Blood Pressure at three months | three months
  Each blood pressure data point was the average of 3 measurements measured 5 minutes apart while seated.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O'Malley, MD, MPH, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Medical Military Center (WRNMMC), Bethesda, Maryland, United States